CLINICAL TRIAL: NCT05229341
Title: Evaluation of DNA Methylation Signatures in Diagnosis and Management of Thyroid Nodules
Brief Title: Evaluation of DNA Methylation Signatures for the Diagnosis and Management of Thyroid Nodules
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21129; NCI-2021-12556 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21129 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2022-02-04; First posted 2022-02-08 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Gland Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Molecular Diagnostic Techniques; Biopsy, Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (needle biopsy, DDMS-2) (Experimental): Patients undergo needle biopsy for collection of tissue samples. Tissue samples are analyzed using DDMS-2. Patients' medical records are also reviewed.
  Interventions: Procedure: Diagnostic Procedure; Other: Electronic Health Record Review; Procedure: Needle Biopsy

INTERVENTIONS:
Procedure: Diagnostic Procedure — Analysis via DDMS-2
  Other Names: Diagnostic Method; Diagnostic Technique; Diagnostic Test
Other: Electronic Health Record Review — Review of medical records
Procedure: Needle Biopsy — Undergo needle biopsy
  Other Names: Aspiration Biopsy; Puncture Biopsy

SUMMARY:
This clinical trial evaluates deoxyribonucleic acid (DNA) methylation signatures in diagnosing and managing thyroid nodules. The purpose of this research is to develop a new test for thyroid cancer. This test will use needle biopsies (small collections of tissue with a needle) from the thyroid to determine whether the participant has a malignant (cancer) or benign (not showing cancer) thyroid tumor. The information learned from this trial may help develop a more accurate test so that patients do not have unnecessary surgeries for nodules that are thought to be suspicious but are actually benign.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of Diagnostic DNA Methylation Signatures (DDMS-2) results (positive predictive value [PPV], negative predictive value [NPV], sensitivity and specificity) on physician decision-making for clinical management of 800 indeterminate thyroid nodules.

SECONDARY OBJECTIVES:

I. To determine sensitivity and specificity, PPV, NPV of DDMS-2 with 1450 needle biopsies including 800 needle biopsies with indeterminate cytopathology.

II. Compare the diagnostic accuracy between DDMS-2 and two currently used diagnostic approaches based on genetic alterations and gene expression within the same prospective cohort of 800 indeterminate needle biopsies.

OUTLINE:

Patients undergo needle biopsy for collection of tissue samples. Tissue samples are analyzed using DDMS-2. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients without impaired decision-making capacity and who are undergoing needle biopsies for thyroid nodule diagnosis
* Over the age of 18
* Any gender, race and ethnicity
* Patients must provide informed consent prior to use of their tissues and clinical data

Exclusion Criteria:

* Children are excluded from the study, since the biology of children thyroid nodules is different from adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1450 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2026-10-22 (Estimated); Study Completion 2026-10-22 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Diagnostic Deoxyribonucleic Acid (DNA) Methylation Signatures (DDMS-2) | Up to 5 years
  The sensitivity of DDMS-2 will be estimated by taking the ratio of the number of true thyroid cancer specimens diagnosed as cancer by DDMS and the total number of thyroid cancer specimens. Will also determine the 95% confidence intervals.
Specificity of DDMS-2 | Up to 5 years
  The specificity will be estimated by taking the ratio of the number of true benign nodules diagnosed as benign by DDMS and the total number of true benign thyroid nodules. Will also determine the 95% confidence intervals.
Positive predictive value (PPV) of DDMS-2 | Up to 5 years
  PPV (number of true thyroid cancer specimens by DDMS / number of thyroid cancers diagnosis by DDMS) will be calculated. Will also determine the 95% confidence intervals.
Negative predictive value (NPV) of DDMS-2 | Up to 5 years
  NPV (number of true benign nodules diagnosed by DDMS/number of benign diagnosis by DDMS) will be calculated. Will also determine the 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: John H Yim, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States